CLINICAL TRIAL: NCT03634527
Title: Auricular Point Acupressure: Examining the Scientific Underpinnings of Pain Relief
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding duration ended.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: IRB00119665
Record Dates: First submitted 2018-03-05; First posted 2018-08-16 (Actual); Last update posted 2021-03-29 (Actual); Status verified 2019-03

CONDITIONS: Chemotherapy-induced Peripheral Neuropathy (CIPN)

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: Participants and outcome assessor will be masked for the treatment that participants received (actual treatment vs sham treatment).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Auricular Point Acupressure (Experimental): Auricular points related to Chemotherapy-induced peripheral neuropathy (CINP) will be used for the intervention.
  Interventions: Behavioral: Auricular Point Acupressure
- Control Auricular Point Acupressure (Sham Comparator): Auricular points not related to CINP will be used for the intervention.
  Interventions: Behavioral: Control Auricular Point Acupressure-

INTERVENTIONS:
Behavioral: Auricular Point Acupressure — Light touch using vaccaria seeds on specific points of the ear
  Arms: Auricular Point Acupressure
Behavioral: Control Auricular Point Acupressure- — Light touch using vaccaria seeds on different points of the ear (compared to the APA group).
  Arms: Control Auricular Point Acupressure

SUMMARY:
Chemotherapy-induced peripheral neuropathy (CIPN)-numbness, burning and stunning pain distributed in hands and feet-is a major challenge among cancer patients. Even after completion of chemotherapy, CIPN persists among ~30-40% of cancer patients, which can negatively impact quality of life. The only drug (duloxetine) better than placebo in a randomized control trial improved pain intensity by 0.72 points on a scale of 0-10, which cannot manage CIPN effectively. A better pain management strategy clearly needs to be developed.

The investigators propose to test auricular point acupressure (APA), a non-invasive, easily administered, patient-controlled, and non-pharmacological strategy, to provide rapid, safe, and effective pain relief so that cancer patients can self-manage their CIPN. APA involves an acupuncture-like stimulation of the ear without needles. With APA, small seeds are taped to specific ear points. The patient is taught to apply pressure to the seeds, with the thumb and index finger, three times a day (morning, noon, and evening) for three minutes each session to achieve pain relief. The investigators have developed a detailed APA protocol to teach health-care providers without experience in acupuncture and traditional Chinese Medicine that investigators can learn about APA in brief educational seminars as a treatment including the systematic identification of ear points (called auricular diagnosis). The investigators teach methods that enable patients to continue using APA to self-manage their pain. However APA is not available in current U.S. health care setting yet.

Quantitative sensory testing (QST) and fMRI in acupuncture have provided new objective methods for measuring pain. QST provides an evaluation of peripheral and central mechanisms of pain by quantifying stimulus-evoked negative and positive sensory phenomena to evaluate a participant's perception of threshold values regarding pain generated through touch (A beta fibers), warmth (C fibers), cold (A delta fibers), and heat (C fibers). Studies have demonstrated changes in heat, pressure, and mechanical pain thresholds immediately following acupuncture; however no study in APA yet. Brain imaging studies in acupuncture indicate that acupuncture can restore normal functional connectivity related to pain reduction. In conjunction with the investigators pilot data demonstrating that APA impacts neural-immune signaling in patients with chronic low back pain, the investigators hypothesize that APA may likewise induce pain relief through the stimulation of A beta fibers and/or C fibers to increase the pain threshold, endogenous opioid binding (releasing inflammatory cytokines), and alter brain networks of central processing in the hypothalamic-pituitary-adrenocortical axis to achieve analgesia.

The investigators plan to study the mechanisms underpinning pain sensitivity and pain processing due to APA on CIPN. Along with the clinical and subjective CIPN outcomes, objective outcomes will include physiological change in pain sensory thresholds (measured by quantitative sensory testing), brain change associated with pain processing (measured by fMRI), and neuro-transmitters (measured by inflammatory cytokines).

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients who are 18 years of age or olde
* Able to read and write English
* Have CIPN due to received neurotoxic chemotherapy for cancer
* Had average intensity of pain due to CIPN ≥ 4 on a 11-point numerical pain scale in the previous week
* Pain > 3 months duration attributed to CIPN.

Exclusion Criteria:

* Use of an investigational agent for pain control concurrently or within the past 30 days;
* Use of an implantable drug delivery systems, e.g. Medtronic Synchromed
* Prior celiac plexus block, or other neurolytic pain control treatment
* Other identified causes of painful paresthesia existing prior to chemotherapy (e.g., radiation or malignant plexopathy, lumbar or cervical radiculopathy, pre-existing peripheral neuropathy of another etiology
* Allergy to latex (the tapes for the APA include latex).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-02-15 (Actual); Primary Completion 2019-01-30 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
Change in Pain intensity as assessed by the Brief Pain Inventory-short form (BPI-sf) questionnaire | Baseline, weekly upto 4 Weeks.
  The Brief Pain Inventory-short form (BPI-sf) questionnaire includes assessment of pain location and multiple aspects of severity of pain, numbness, tingling, and stiffness, including worst, least, average pain, and present, as well as the interference with daily activities. The Brief Pain Inventory-short form (BPI-sf) has a total score ranging from 0 to 10 with higher scores indicating more pain.

SECONDARY OUTCOMES:
Change in Quantitative Sensory Testing (QST) score | Baseline, weekly upto 4 weeks
  Quantitative Sensory Testing will be measured by cold pressor testing, conditional pain modulation, mechanical pain threshold. The percentage of change score (from each end point to baseline) will be used (0-100) with higher scores indicating less pain
Change in pain response assessed by functional MRI Scan | baseline, post-4weekly APA treatment, and one month followup
  The baseline rs-fMRI will be performed, followed by 10 min of APA. Immediately after the treatment, a repeat fMRI will then be performed. All MRIs will be acquired on a 3.0 Tesla Siemens Trio Tim system (Siemens Medical Solutions, Erlangen, Germany) using a 12-channel head matrix coil T2*-weighted bold functional images covering entire cerebrum and cerebellum. fMRI will take ~45 minutes. The imaging data will be processed using Statistical Parametric Mapping version 8.
Change in functional status as assessed by the e Patient-Reported Outcomes Measurement Information System (PROMIS) 29 scale | weekly up to one month post-intervention
  PROMIS 29 will be used to assess Anxiety, Depression, Fatigue, and Sleep Disturbance.The PROMIS-29 scale, which includes: Pain Interference - 4 items; Pain Intensity- 1 item; Physical Function - 4 items; Fatigue - 4 items;Depression - 4 items; Anxiety - 4 items; Sleep Disturbance - 4 items; Satisfaction with Social Participation- 4 items
Change in Inflammatory Cytokines | baselines, weekly upto 4 weeks
  It will be measured by blood serum

CONTACTS AND LOCATIONS:
Overall Officials: Chao Hsing Yeh, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
Have not decided since this is a pilot study.